CLINICAL TRIAL: NCT05835388
Title: The South Texas Aging Registry and Repository (STARR)
Brief Title: The South Texas Aging Registry and Repository
Acronym: STARR
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Other Study IDs: HSC20150610H
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Aging
Keywords: Older adults; Genetic material; Biorepository

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and serum will be stored for future research after obtaining blood sugar level, and other measures such as lipids, liver and kidney function.
  Genetic material will be obtained from blood to provide the biology of aging and aging-related disorders.
  Fat samples collected from a biopsy for future genetic research. Skin tissue will be collected by a punch biopsy for future genetic research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Study: Community dwelling adults from the South Texas area who are interested in volunteering for research studies on aging. This will facilitate the inclusion of older adults and minority in research studies and help to increase the quantity and quality of research relating to them.
- KAPP Sen Tissue Mapping Study: The substudy KAPP Sen TMC will enroll eligible STARR participants to undergo repeat assessments over two years. KAPP Sen TMC is a collaborative effort between UT Health San Antonio, Jackson Laboratory for Genomic Medicine (JAX-GM), Brigham and Women's Hospital, Joslin Diabetes Center, UConn Health Center on Aging and Mayo Clinic to characterize cellular senescence in terms of its presence and heterogeneity in healthy human tissues, as well as its tissue burden, spatial distribution, and biological features in a diverse study population.

SUMMARY:
This research registry and repository was designed because the investigators want to learn about how to improve the health and quality of life of older adults.

DETAILED DESCRIPTION:
The South Texas Aging Registry and Repository (STARR) is a database and specimen resource of community dwelling adults from the South Texas area who are interested in volunteering for research studies on aging. The goal is to assist in the inclusion of older adults in clinical research studies and to help to increase the quantity and quality of research relating to them. This registry and repository can be used for various purposes ranging from describing the natural history of aging, identifying risk factors for premature aging, and the real-world effectiveness of life-extending therapies. Collection and storage of biological samples and patient-reported data from of Individuals can help advance research and the development of new awareness of basic mechanisms that play a part in healthy aging or premature death.

ELIGIBILITY:
Inclusion Criteria STARR:

-Age 18 years or older

Inclusion Criteria KAPP Sen TMC:

-Age 20 years and older

Exclusion Criteria STARR:

* Inability to provide informed consent
* Pregnancy

Exclusion Criteria KAPP Sen Tissue Mapping Center (TMC) Study:

* Diabetes
* Hypertension with end-organ damage
* BMI>30
* GFR<60 ml/min/1.73 m2
* Cardiovascular disease
* Pancreatitis
* Malignancy other than non-melanoma skin cancers
* Active, uncontrolled pulmonary, hepatic, infectious, gastrointestinal, endocrine, neurologic, or inflammatory disease.
* Chronic use of systemic steroids or use of agents with senolytic activity
* Any disease or condition considered to be exclusionary based on the clinical option and discretion of PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling adults from the South Texas area who are interested in volunteering for research studies on aging.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Collection of STARR repository data | Baseline to one day
  De-identified repository data and samples will be made available to outside investigators for future studies related to aging

SECONDARY OUTCOMES:
KAPP Sen TMC repository data | Baseline to one year
  Eligible STARR participants to undergo repeat assessments to characterize cellular senescence

CONTACTS AND LOCATIONS:
Overall Officials: Sara Espinoza, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
New prospective studies and those involving interacting with human subjects: Participants/research volunteers who agree to be re-contacted will be matched with future studies which they are likely to qualify for based upon information provided by each STARR participant at the time of enrollment and which is gathered using provided samples.
  KAPP Sen TMC will support the use of a web-based platform to connect and facilitate entering, sharing, and exchanging data among collaborates. Data will be exported to a web portal developed in conjunction with the CODCC where the research community can request access to molecular data and corresponding biospecimen data, such as clinical, demographic, and biospecimen handling data.
Supporting Information: Study Protocol, SAP
Time Frame: Requests from investigators to obtain data/specimens from the repository must be submitted in writing using an official repository request form, along with study protocol and documentation of appropriate approvals. Requests will be reviewed on a monthly basis by members of the Repository Executive Committee. Request to access data or specimens will be processed and entered into the Repository Log by the Repository Coordinator and submitted for review by the Executive Committee each month.